CLINICAL TRIAL: NCT01195155
Title: Transcriptomic Profile of Subcutaneous Adipose Tissue of Young Women With PCOS Followin 6 Weeks Supplementation With n-3 PUFA Versus Olive Oil Placebo
Brief Title: Transcriptomic Profile of Adipose Tissue Following n-3 Polyunsaturated Fatty Acid (PUFA) Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Adelaide and Meath Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Dr James Gibney, The Adelaide and Meath Hospital Incorporating the National Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DDC-UCD-ATN3
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2008-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LC n-3 PUFA (Active Comparator): Supplementation with 4 x 1g fish oil capsules (Seven Seas, Ireland) containing 1.9g combined EPA and DHA daily for 6 weeks.
  Interventions: Dietary Supplement: LC n-3 PUFA (fish oil) Supplement
- Placebo (olive oil) supplement (Placebo Comparator): 4 x 1g olive oil capsules (Millas Inc) were given daily for 6 weeks.
  Interventions: Dietary Supplement: LC n-3 PUFA (fish oil) Supplement
- Wash out period (No Intervention): A 6 week wash out period separated the LC n-3 PUFA and the Placebo (olive oil) arms. During this period the subjects took no supplements. This arm was designed to minimise a cross-over effect.
  Interventions: Dietary Supplement: LC n-3 PUFA (fish oil) Supplement

INTERVENTIONS:
Dietary Supplement: LC n-3 PUFA (fish oil) Supplement — 4 x 1g LC n-3 PUFA (fish oil)supplement containing 1.9g EPA and DHA given daily for 6 weeks
  Other Names: LC n-3 PUFA (fish oil); Placebo (PL); Wash-out (WO)

SUMMARY:
Adipose tissue is a central organ involved in mediating metabolic health, and so the investigation of treatments which improve adipose tissue function is warranted. LC n-3 polyunsaturated fatty acid (PUFA) have been shown to exert positive effects on adipose tissue gene expression in previous studies. However this has not been investigated in women with polycystic ovary syndrome (PCOS), a population shown to display a degree of adipose tissue dysfunction. The aim of this study was to determine the impact of LC n-3 PUFA supplementation on gene expression profiles of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Had a positive diagnosis of PCOS as defined according to the NIH criteria as chronic oligomenorrhoea (< 9 menstrual cycles per year) and clinical and/or biochemical evidence of hyperandrogenism, in the absence of other disorders causing the same phenotype. Clinical criteria included hirsutism with a Ferriman-Galwey score greater than 9, acne or male pattern alopecia; biochemical criteria included total-testosterone, androstenedione or dehydroepiandrosterone sulphate (DHEAS) greater than the laboratory reference range.
* Were between the ages of 18 and 40

Exclusion Criteria:

* Were under 18 years or greater than 40 years old,
* Were non-Caucasian
* Were pregnant, lactating or trying to conceive
* Had a body mass index (BMI) <18kg/m2 or >50kg/m2
* Had a recent illness or any chronic illness likely to influence results
* Were taking any medications likely to influence the results including hormonal contraception, antihypertensives, lipid lowering medications, antiplatelet agents, anti-inflammatory agents
* Were taking nutritional supplements
* Consumed greater than 2 portions of oily fish per week

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Gene expression profiling subcutaneous adipose tissue of young women with PCOS following LC n-3 PUFA supplementation versus control | Following 6 weeks of LC n-3 PUFA supplementation versus 6 weeks olive oil placebo supplementation
  Gene expression profiles were assessed by mircoarray analysis from samples of subcutaneous adipose tissue obtained from subjects following LC n-3 PUFA and placebo supplementation. Single gene changes and pathway analyses will be conducted to assess potential differences between PCOS and control samples.

SECONDARY OUTCOMES:
Assessment of biomarkers of hormonal and metabolic health in young women with PCOS following LC n-3 PUFA supplementation versus placebo | Following 6 weeks of LC n-3 PUFA supplementation versus 6 weeks olive oil placebo supplementation
  Key biomarkers of metabolic health (plasma lipid profile, inflammatory markers and adipokines) and androgenic hormonal profile (testosterone, androstenedione, DHEAS) were assessed by measuring circulating concentrations in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: James Gibney, Dr, Principal Investigator — The Adelaide and Meath Hospital; Helen M Roche, Prof, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - The Adelaide and Meath Hosptial, Dublin, Leinster
  - Nutrigenomics Group, University College Dublin, Dublin, Leinster